CLINICAL TRIAL: NCT01356173
Title: An Open-Label, Phase I, Dose Escalation Study Evaluating the Safety and Tolerability of GDC-0349 in Patients With Locally Advanced or Metastatic Solid Tumors or Non Hodgkin's Lymphoma
Brief Title: Evaluating the Safety and Tolerability of GDC-0349 in Patients With Locally Advanced or Metastatic Solid Tumors or Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKI4956g; MP00807 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma, Solid Tumor
Keywords: solid cancers
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — GDC-0349

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0349

INTERVENTIONS:
Drug: GDC-0349 — Oral escalating dose

SUMMARY:
This is an open-label, multicenter, Phase I, dose-escalation study to assess the safety, tolerability, and pharmacokinetic (PK) of GDC-0349 administered once daily (QD), orally (PO).

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, locally advanced or metastatic solid malignancy or NHL without leukemic phase that has progressed or failed to respond to at least one prior regimen and/or are not candidates for regimens known to provide clinical benefit
* Evaluable or measurable disease per RECIST v1.1 or IWG response criteria for patients with NHL and/or the following: prostate cancer patients with non-measurable disease are eligible if they have two rising prostate-specific antigen (PSA) levels >= 5 ng/mL measured >= 2 weeks apart that meet the PSA, and Working Group criteria for progression prior to initiation of study treatment, and ovarian cancer patients with non-measurable disease are eligible if they have two rising CA-125 levels greater than the ULN >= 2 weeks apart prior to initiation of study treatment.
* ECOG performance status of 0 or 1 at screening
* Life expectancy of >= 12 weeks
* Adequate hematologic and organ function within 14 days prior to initiation of study treatment
* Documented willingness to use an effective means of contraception for both men and women while participating in the study and for 90 days after the last dose of GDC-0349
* Willingness to provide archival tumor tissue

Exclusion Criteria:

* Leptomeningeal disease as the only manifestation of the current malignancy
* History of Type 1 or 2 diabetes requiring daily medication
* Known untreated central nervous system (CNS) malignancies or treated brain metastases that are not radiographically stable for >= 3 months prior to initiation of study treatment
* Active congestive heart failure or ventricular arrhythmia requiring medication
* Uncontrolled ascites requiring weekly large-volume paracentesis for 3 consecutive weeks prior to initiation of study treatment
* Active infection requiring intravenous (IV) antibiotics
* Patients requiring any daily supplemental oxygen
* Uncontrolled hypomagnesemia or hypokalemia
* Any condition requiring anti-coagulants such as warfarin, heparin, or anti-thrombotics. Prophylactic anti-coagulation and/or local application of thrombolytic agents for catheter patency may be allowed for patients with normal INR and with prior approval from the Medical Monitor
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus (HIV) infection
* Any other diseases, active or uncontrolled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or renders the patients at high risk from treatment complications
* Significant traumatic injury within 3 weeks prior to initiation of GDC-0349
* Major surgical procedure within 4 weeks prior to initiation of GDC-0349
* Treatment with chemotherapy, hormonal therapy (except GnRH agonists or antagonists for prostate cancer), immunotherapy, biologic therapy, or radiation therapy (except palliative radiation to bony metastases) as cancer therapy within 4 weeks prior to initiation of study treatment. Kinase inhibitors, approved by national regulatory authorities, may be used up to 2 weeks prior to initiation of GDC-0349, provided that any drug-related toxicity has completely resolved and prior approval is obtained from the Medical Monitor.
* Palliative radiation to bony metastases within 2 weeks prior to initiation of GDC-0349
* Treatment with an investigational agent within 4 weeks prior to initiation of GDC-0349
* Unresolved toxicity from prior therapy, except for alopecia and Grade 1 peripheral neuropathy
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) by NCI CTCAE v4.0 grade and associated dose of GDC-0349 | Up to 30 days

SECONDARY OUTCOMES:
Incidence of adverse events by NCI CTCAE v4.0 grade and associated dose of GDC-0349 | Up to 2 years
Incidence of Grade 3 and 4 abnormalities in safety related laboratory parameters and associated dose of GDC-0349 | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holden, M.D., Study Director — Genentech, Inc.
Locations (2):
- Scottsdale, Arizona, United States
- Toronto, Ontario, Canada